CLINICAL TRIAL: NCT00003474
Title: Phase II Study of Antineoplastons A10 and AS2-1 in Adult Patients With Glioblastoma Multiforme
Brief Title: Antineoplaston Therapy in Treating Adults With Residual/Recurrent/Progressive Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066511; BRI-BT-20 (Other: Burzynski Research Institute)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Glioblastoma Multiforme of the Brain
Keywords: adult glioblastoma; recurrent glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- Antineoplaston therapy (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Adults with a residual/recurrent/progressive Glioblastoma Multiforme will receive Antineoplaston therapy (Atengenal + Astugenal).
  The daily doses of A10 and AS2-1 are divided into six infusions, which are given at 4-hourly intervals. Each infusion starts with infusion of A10 and is immediately followed by infusion of AS2-1.
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)

SUMMARY:
RATIONALE: Current therapies for Glioblastoma Multiforme provide very limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of brain tumors.

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on adults (≥ 18 years of age) with residual/recurrent/progressive Glioblastoma Multiforme.

DETAILED DESCRIPTION:
OVERVIEW: This is a single arm, open-label study in which adults (≥ 18 years of age) with residual/recurrent/progressed Glioblastoma Multiforme receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues for at least 12 months in the absence of disease progression or unacceptable toxicity.

OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in adults (≥ 18 years of age) with residual/recurrent/progressive Glioblastoma Multiforme following initial therapy, including radiotherapy, as measured by an objective response to therapy (complete response, partial response or stable disease).
* To determine the safety and tolerance of Antineoplaston therapy in adults (≥ 18 years of age) with residual/recurrent/progressive Glioblastoma Multiforme.
* To determine objective response, tumor size is measured utilizing MRI scans, which are performed every 8 weeks for the first two years, every 3 months for the third and fourth years, every 6 months for the 5th and sixth years, and annually thereafter.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued to this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed incurable glioblastoma multiforme that has progressed, recurred, or persisted following completion of initial standard therapy (including radiotherapy and/or chemotherapy)

  * Measurable disease by MRI or CT scan
* Brain stem tumor is excluded
* Tumor must be at least 5 mm

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* WBC at least 2,000/mm3
* Platelet count at least 50,000/mm3

Hepatic:

* No liver failure
* Bilirubin no greater than 2.5 mg/dL
* SGOT/SGPT no greater than 5 times upper limit

Renal:

* No history of renal conditions that contraindicate high dosages of sodium
* Creatinine no greater than 2.5 mg/dL

Cardiovascular:

* No uncontrolled hypertension
* No history of congestive heart failure
* No other cardiovascular conditions that contraindicate high dosages of sodium

Pulmonary:

* No serious lung disease (e.g., severe COPD)

Other:

* Not pregnant or nursing
* Fertile patients must use adequate contraception during and for 4 weeks after study
* No active infection
* No other serious medical or psychiatric conditions

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since immunotherapy
* No concurrent immunomodulating agents

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since chemotherapy (unless radiologically proven progression)
* At least 6 weeks since nitrosoureas

Endocrine therapy:

* Corticosteroids allowed

Radiotherapy:

* See Disease Characteristics
* At least 8 weeks since radiotherapy (unless radiologically proven progression)

Surgery:

* Recovered from prior surgery

Other:

* No prior antineoplaston therapy
* Prior cytodifferentiating agent allowed

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 1996-03-14 (Actual); Primary Completion 2003-06-21 (Actual); Study Completion 2003-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty patients were recruited between March 1996 and April 2003. All study subjects were seen at the Burzynski Clinic in Houston TX
Groups:
- Antineoplaston Therapy: Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Antineoplaston therapy (Atengenal + Astugenal): Adults with a residual/recurrent/progressive Glioblastoma Multiforme will receive Antineoplaston therapy (Atengenal + Astugenal).
  The daily doses of A10 and AS2-1 are divided into six infusions, which are given at 4-hourly intervals. Each infusion starts with infusion of A10 and is immediately followed by infusion of AS2-1.
Period: Overall Study
Arm/Group | Antineoplaston Therapy
Started | 40
Completed | 26
Not Completed | 14
Not completed — Not Evaluable | 14

BASELINE CHARACTERISTICS:
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: Years] | 48.8 [26.7 to 71.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response
Description: Objective response rate per Response Assessment in Neuro-Oncology (RANO) for target lesions and assessed by MRI: Complete Response (CR), disappearance of all disease sustained for at least four weeks; Partial Response (PR), >=50% decrease in the sum of the products of of the greatest perpendicular diameters of all measurable enhancing lesions, sustained for at least four weeks.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 26
Participants
  Complete Response | 1
  Partial Response | 1
  Stable Disease | 5
  Progressive Disease | 19

2. Secondary Outcome: Percentage of Participants Who Survived
Description: 6 months, 12 months, 24 months, 36 months, 48 months, 60 months overall survival
Time Frame: 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
Population: All study subjects receiving any Antineoplaston therapy
Measure: Number; unit: Percentage of participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 40
Percentage of participants
  6 months overall survival | 45.0
  12 months overall survival | 22.5
  24 months overall survival | 2.5
  36 months overall survival | 2.5
  48 months overall survival | 2.5
  60 months overall survival | 2.5

ADVERSE EVENTS:
Time Frame: 7 years, 3 months
Description: Forty patients were recruited between March 1996 and June 2003. All study subjects were seen at the Burzynski Clinic in Houston TX
Arm/Group | Antineoplaston Therapy
Serious Adverse Events (participants affected / at risk) | 17/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=40)
Hemoglobin (Blood and lymphatic system disorders) | 1 — The Hemoglobin was not related to Antineoplaston therapy.
Hypertension (Cardiac disorders) | 1 — The Hypertension was not related to Antineoplaston Therapy.
Central Venous Catheter Infection (General disorders) | 3 — The Central Venous Catheter Infections were not related to Antineoplaston Therapy
Dehydration (Gastrointestinal disorders) | 1 — The Dehydration was not related to Antineoplaston Therapy.
Vomiting (Gastrointestinal disorders) | 1 — The Vomiting was not related to Antineoplaston Therapy.
Infection (documented clinically): Bladder (urinary) (Infections and infestations) | 1 — The Infection (documented clinically): Bladder (urinary) was not related to Antineoplaston Therapy.
Infection (documented clinically): Lung (pneumonia) (Respiratory, thoracic and mediastinal disorders) | 2 — The Infections (documented clinically): Lung (pneumonias) were not related to Antineoplaston Therapy
Muscle weakness: Whole body/generalized (Musculoskeletal and connective tissue disorders) | 1 — The Muscle weakness: Whole body/generalized was not related to Antineoplaston Therapy
Seizure (Nervous system disorders) | 3 — The Seizures were not related to Antineoplaston Therapy.
Somnolence/depressed level of consciousness (Nervous system disorders) | 3 — The Somnolences/depressed levels of consciousness were not related to Antineoplaston Therapy.
Syncope (fainting) (Nervous system disorders) | 2 — The Syncopes (faintings) were not related to Antineoplaston Therapy.
Pain: Head/headache (Nervous system disorders) | 2 — The Pain: Head/headaches were not related to Antineoplaston Therapy.
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 — The Dyspneas (shortnesses of breath) were not related to Antineoplaston Therapy.
Thrombosis/thrombus/embolism (Vascular disorders) | 1 — The Thrombosis/thrombus/embolism was not related to Antineoplaston Therapy.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=40)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 7
Tinnitus (Ear and labyrinth disorders) | 3
Hemoglobin (Blood and lymphatic system disorders) | 7
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 4
Lymphopenia (Blood and lymphatic system disorders) | 8
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 3
Platelets (Blood and lymphatic system disorders) | 5
Supraventricular and nodal arrhythmia: Sinus bradycardia (Cardiac disorders) | 2
Hypertension (Cardiac disorders) | 5
Hypotension (Cardiac disorders) | 2
Central Venous Catheter: Infection (Infections and infestations) | 5
Central Venous Catheter: Non-functional (General disorders) | 12
Central Venous Catheter: Other (General disorders) | 2
Central Venous Catheter: Thrombosis/embolism (General disorders) | 3
Constitutional Symptoms - Other (General disorders) | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 23
Insomnia (General disorders) | 4
Weight gain (General disorders) | 3
Fever (General disorders) | 3
Edema (General disorders) | 21
Cushingoid appearance (Endocrine disorders) | 2
Anorexia (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 5
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 15
Vomiting (Gastrointestinal disorders) | 11
Hemorrhage, GU: Urinary NOS (Renal and urinary disorders) | 4
Infection (documented clinically): Bladder (urinary) (Infections and infestations) | 4
Infection (documented clinically): Blood (Infections and infestations) | 2
Infection (documented clinically): Lung (pneumonia) (Infections and infestations) | 4
Infection (documented clinically): Mucosa (Infections and infestations) | 3
Infection (documented clinically): Sinus (Infections and infestations) | 2
Infection (documented clinically): Upper airway NOS (Infections and infestations) | 2
Infection (documented clinically): Urinary tract NOS (Infections and infestations) | 3
Infection: Lung (pneumonia) (Infections and infestations) | 2
Infection: Mucosa (Infections and infestations) | 2
Infection: Opportunistic infection (Infections and infestations) | 5
Albumin, serum-low (hypoalbuminemia) (Investigations) | 3
Alkaline phosphatase (Investigations) | 2
GGT (gamma-Glutamyl transpeptidase) (Investigations) | 3
Hypercholesteremia (Investigations) | 4
Hyperglycemia (Investigations) | 12
Hypernatremia (Investigations) | 25
Hypertriglyceridemia (Investigations) | 3
Hypocalcemia (Investigations) | 3
Hypoglycemia (Investigations) | 7
Hypokalemia (Investigations) | 34
Hypomagnesemia (Investigations) | 3
Hyponatremia (Investigations) | 2
Proteinuria (Investigations) | 5
SGOT (Investigations) | 6
SGPT (Investigations) | 8
Ataxia (incoordination) (Nervous system disorders) | 4
Confusion (Nervous system disorders) | 19
Dizziness (Nervous system disorders) | 15
Memory impairment (Nervous system disorders) | 2
Mood alteration: Agitation (Nervous system disorders) | 2
Mood alteration: Anxiety (Nervous system disorders) | 2
Mood alteration: Depression (Nervous system disorders) | 4
Neuropathy: motor (Nervous system disorders) | 6
Psychosis (hallucinations/delusions) (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 13
Somnolence/depressed level of consciousness (Nervous system disorders) | 22
Speech impairment (Nervous system disorders) | 5
Syncope (fainting) (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 3
Diplopia (Nervous system disorders) | 2
Ophthalmoplegia/diplopia (double vision) (Nervous system disorders) | 2
Vision-blurred vision (Nervous system disorders) | 2
Pain: Back (Musculoskeletal and connective tissue disorders) | 2
Pain: Head/headache (Nervous system disorders) | 15
Pain: Joint (Musculoskeletal and connective tissue disorders) | 3
Pain: Muscle (Nervous system disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 9
Incontinence, urinary (Renal and urinary disorders) | 3
Urinary frequency/urgency (Renal and urinary disorders) | 2
Thrombosis/thrombus/embolism (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No